CLINICAL TRIAL: NCT05951829
Title: Effects of Action Observation Therapy and Mirror Therapy on Upper Extremity Functions in Children With Unilateral Cerebral Palsy: A Randomized Controlled Study With 1 Month Follow-Up
Brief Title: Effects of Action Observation Therapy and Mirror Therapy in Children With Unilateral Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SEDANUR GÜRLEK, Hacettepe University-Principal Investigator-PhD Student, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG13
Record Dates: First submitted 2023-06-21; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Cerebral Palsy; Functioning; Upper Extremity Problem
MeSH Terms: conditions — Cerebral Palsy | interventions — Mirror Movement Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cerebral Palsy (Other)
  Interventions: Other: Action Observation Therapy

INTERVENTIONS:
Other: Action Observation Therapy — Action Observation Therapy Mirror Therapy
  Other Names: Mirror Therapy

SUMMARY:
The aim of this study was to examine the effects of action observation therapy and mirror therapy on upper extremity functions in children with unilateral cerebral palsy. In the study, the 1st group is the Action Observation Therapy group and will receive 18 sessions of practice. The second group is the mirror therapy group and will receive a total of 18 practice sessions. To evaluate the outcome measures of children's upper extremity functions; Canadian Occupational Performance Mesure (COPM), Goal Achievement Scale (GAS), Shriners Hospital Upper Extremity Function Scale (SHUEE), Melbourne Unilateral Upper Extremity Function Evaluation Test and ABILHAND Questionnaire will be used. The satisfaction of the families with the therapy process will be evaluated with the Visual Analog Scale (VAS).

DETAILED DESCRIPTION:
The aim of this study was to examine the effects of action observation therapy and mirror therapy on upper extremity functions in children with unilateral cerebral palsy. In the study, the 1st group is the Action Observation Therapy group and will receive 18 sessions of practice. The second group is the mirror therapy group and will receive a total of 18 practice sessions. To evaluate the outcome measures of children's upper extremity functions; Canadian Occupational Performance Mesure (COPM), Goal Achievement Scale (GAS), Shriners Hospital Upper Extremity Function Scale (SHUEE), Melbourne Unilateral Upper Extremity Function Evaluation Test and ABILHAND Questionnaire will be used. The satisfaction of the families with the therapy process will be evaluated with the Visual Analog Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 5 and 15
* Being diagnosed with unilateral cerebral palsy
* Be in one of the levels 1,2 and 3 according to the MACS dexterity classification
* Upper extremity Modified Ashworth Scale score less than or equal to 2 attending primary school

Exclusion Criteria:

* Having a visual impairment recorded in the health report
* To have any neurological, orthopedic, and psychiatric diagnosis in addition to the diagnosis of cerebral palsy
* Difficulty understanding and applying verbal and visual commands
* To have undergone any surgical intervention or botox in the last 3 months

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-07-10 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
The Canadian Occupational Performance Measure | 6 weeks
  Assessment
Goal Attainment Scaling | 6 weeks
  Assessment
Shriners Hospital Upper Extremity Evaluation | 6 weeks
  Assessment
Melbourne Assessment of Unilateral Upper Limb Function | 6 weeks
  Assessment
ABILHAND-Kids Questionnaire | 6 weeks
  Assessment
Visual Analogue Scale | 6 weeks
  Assessment